CLINICAL TRIAL: NCT04157569
Title: Monitoring Circulating Tumor DNA After Chemotherapy in Elderly Patients With Acute Leukemia
Brief Title: CtDNA After Chemotherapy in Elderly Patients With Acute Leukemia
Status: Recruiting | Type: Observational
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Principal Investigator, Navy General Hospital, Beijing
Other Study IDs: NavyGHB-006
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venipuncture peripheral blood bone marrow finger stick peripheral blood saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will monitor CtDNA After Chemotherapy in Elderly Patients With AL

DETAILED DESCRIPTION:
This study will use droplet digital PCR (ddPCR) method to quantify peripheral blood plasma mutant allele frequency (MAF) in elderly acute leukemia patients after chemotherapy to evaluate the clinical value of CtDNA .

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male
* not pregnant female
* patients >=60 years old
* Diagnosis of acute leukemia

Exclusion Criteria:

* Pregnancy
* HIV positive
* patients >=100 years old

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population include old AML patients with somatic mutations
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of relapse(CIR) | through study completion, an average of 1 year
  cumulative incidence of relapse

SECONDARY OUTCOMES:
overall survival (OS) | through study completion, an average of 2 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, MD, Study Chair — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, China